CLINICAL TRIAL: NCT01804595
Title: A Randomized Control Trial of Sun Protection Interventions for Operating Engineers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Sonia Duffy, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N015454-00
Record Dates: First submitted 2013-02-26; First posted 2013-03-05 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Skin Cancer Prevention
Keywords: Worksite intervention; Sun protection intervention; Operating Engineers
MeSH Terms: interventions — Sunscreening Agents; Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sunscreen (Experimental): To reduce barriers to obtaining sunscreen and serve as cues to action, this group will be mailed during the months of May through September, a supply of SPF30 sunscreen lotion (known to prevent sun burning and skin cancer). The mailing will consist of large bottles of sunscreen and a small bottle that can be refilled and attached to their huge key rings that hang off of their belts.
  Interventions: Other: Sunscreen; Behavioral: Education
- Text Message Reminders (Experimental): As cues to action, this group will receive 60 cellular telephone text-messages on three random mornings per week during the month of May, June, July, August, and September when UV rays are the highest. Using an internet text-messaging service, the messages will be computer generated and sent to Operating Engineers and contain information about weather conditions and various reminders (e.g., "Put on sunscreen today" or "Wow, it's a hot one, you know what to do!").
  Interventions: Behavioral: Text-Message Reminders; Behavioral: Education
- Sunscreen and Text Message Reminders (Experimental): Just as multimodal interventions such as surgery and radiation can be used to treat skin cancer, multimodal behavioral interventions may reduce sun burning and prevent skin cancer. To determine if the combination of these interventional components results in improvements above and beyond the individual parts, both sunscreen and text messaging interventions will be provided in addition to education.
  Interventions: Other: Sunscreen; Behavioral: Text-Message Reminders; Other: Sunscreen and Text Message Reminders; Behavioral: Education
- Education (Active Comparator): A 30-minute, picture enhanced power point presentation will be offered to all Operating Engineers during their annual safety trainings. The content of the power point presentation will include information on incidence and prevalence of skin cancer especially among outdoor workers, types of skin cancers and skin cancer risk, sunburn, Sun Protection Factor (SPF), sun protection behaviors including sunscreen use, correct application of sunscreen, types of products, and the new Food and Drug Administration (FDA) labeling of sunscreen products. In addition, other sun protection behaviors such as wearing hats, sunglasses, using shade, etc., will be discussed.
  Interventions: Behavioral: Education

INTERVENTIONS:
Other: Sunscreen
  Arms: Sunscreen; Sunscreen and Text Message Reminders
Behavioral: Text-Message Reminders
  Arms: Sunscreen and Text Message Reminders; Text Message Reminders
Other: Sunscreen and Text Message Reminders
  Arms: Sunscreen and Text Message Reminders
Behavioral: Education

SUMMARY:
This is a randomized controlled trial testing the efficacy of 4 sun protection interventions--education only; education and mailed sunscreen; education and text message reminders; and education, mailed sunscreen, and text message reminders--among Michigan Operating Engineers. Pre- and post-intervention surveys will be collected to determine changes in sunscreen use and sun burning, the primary outcome variables. The investigators hypothesize that all interventions will increase sunscreen use and reduce burning and that the education-only intervention will have the least effect of the 4 interventions while the education, mailed sunscreen, and text messaging arm will have the greatest effect.

DETAILED DESCRIPTION:
The education intervention will be provided during regularly scheduled safety training sessions, and the text messages and mailed sun screen (SPF30)interventions will be offered during the summer when UV rays are at their highest. Inclusion criteria are Operating Engineers who:1)are greater than 18 years of age; 2) are interested in enrolling in the sun protection study; 3) own a cell-phone that accepts text messages; and 4) are willing to share their phone number with the study team. Based on power analysis, 256 subjects are needed to have 80% power to detect medium sized effects on primary outcomes. Accounting for a 20% attrition rate, 320 subjects will be recruited. The analyses will include: a) paired t-tests to determine changes over time (from pre-intervention to post-intervention) in outcome variables (sunscreen use and burning) separately in the 4 intervention groups, b) Repeated Measures Analysis of Variance (RM-ANOVA) to compare the changes in outcomes across the 4 groups, and c) t-tests on change scores as follow-ups to the RM-ANOVA to determine exactly which groups differ from each other. Sub-analyses will explore if particular subgroups of Operating Engineers (e.g., demographic, heath behavior, and job type subgroups) differ in sunscreen use and sun burning pre-and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years of age
* interested in enrolling in the sun protection study
* owning a cell-phone that accepts text messages
* willing to share their phone number with the study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Sunscreen use | Baseline
  Subjects will complete a baseline survey during safety training sessions in Winter when they get the educational intervention. In the past summer, on the days when you were outside in the sunlight, how often did you use sun block (never, some of the time, about half the time, most of the time, always)?
Sun Burning | Baseline
  Subjects will complete a baseline survey during safety training sessions in Winter when they get the educational intervention. On average, how many times did you get a sunburn this past summer (0, 1, 2, 3, 4 or more times)?
Sunscreen use | Post-intervention
  Subjects will be texted or phoned this question monthly during the intervention period and will again receive this question on the longer follow up survey up to 5 months after the interventions end. In the past summer, on the days when you were outside in the sunlight, how often did you use sun block (never, some of the time, about half the time, most of the time, always)?
Sun Burning | Post-intervention
  Subjects will be texted or phoned this question monthly during the intervention period and will again receive this question on the longer follow up survey up to 5 months after the interventions end. On average, how many times did you get a sunburn this past summer(0, 1, 2, 3, 4 or more times)?

CONTACTS AND LOCATIONS:
Overall Officials: Sonia A Duffy, PhD, RN, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Nursing, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Walkosz BJ, Buller DB, Andersen PA, Scott MD, Dignan MB, Cutter GR, Maloy JA. Increasing sun protection in winter outdoor recreation a theory-based health communication program. Am J Prev Med. 2008 Jun;34(6):502-9. doi: 10.1016/j.amepre.2008.02.011. PMID 18471586
- [Background] Armstrong AW, Watson AJ, Makredes M, Frangos JE, Kimball AB, Kvedar JC. Text-message reminders to improve sunscreen use: a randomized, controlled trial using electronic monitoring. Arch Dermatol. 2009 Nov;145(11):1230-6. doi: 10.1001/archdermatol.2009.269. PMID 19917951
- [Derived] Duffy SA, Ronis DL, Waltje AH, Choi SH. Protocol of a randomized controlled trial of sun protection interventions for operating engineers. BMC Public Health. 2013 Mar 26;13:273. doi: 10.1186/1471-2458-13-273. PMID 23530608
- See also: FDA announces new requirements for over-the-counter (OTC) sunscreen products marketed in the U.S. 2011 — http://www.fda.gov/drugs/resourcesforyou/consumers/buyingusingmedicinesafely/understandingover-the-countermedicines/ucm258468.htm